CLINICAL TRIAL: NCT00944814
Title: Assessment of the Acceptability of Zinc-fortified Lipid Based Nutrient (LNS) Prepared for Young Burkinabe Children
Brief Title: Acceptability of Zinc-fortified Lipid-based Nutrient Supplements
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Collaborators: Université Polytechnique de Bobo-Dioulasso (Other); Helen Keller International (Other); Bill and Melinda Gates Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 200917273; iLiNS-ACCEPT-Zinc
Record Dates: First submitted 2009-07-21; First posted 2009-07-23 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Malnutrition
Keywords: Lipid-based nutrient supplement; Prevention of malnutrition; Prevention of micronutrient deficiencies; Zinc
MeSH Terms: conditions — Malnutrition | interventions — Hypoxanthine Phosphoribosyltransferase; Zinc

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LNS with zinc (Experimental): LNS containing 10 mg zinc per 20 g dose of LNS
  Interventions: Dietary Supplement: LNS with zinc
- LNS without zinc (Placebo Comparator): LNS containing no zinc
  Interventions: Dietary Supplement: LNS without zinc

INTERVENTIONS:
Dietary Supplement: LNS with zinc — Lipid-based nutrient supplement (LNS) containing 10 mg zinc/20 g LNS dose
  Other Names: Nutriset lipid-based nutrient supplement with zinc
  Arms: LNS with zinc
Dietary Supplement: LNS without zinc — LNS containing no zinc
  Other Names: Nutriset lipid-based nutrient supplement without zinc
  Arms: LNS without zinc

SUMMARY:
The purpose of the study is to assess the acceptability of the two lipid-based nutrient supplement (LNS) formulations containing no zinc and a high amount of zinc (10 mg zinc / 20 g dose of LNS). The hypothesis is that both products will be equally accepted by children and mothers.

DETAILED DESCRIPTION:
We plan to conduct a series of acceptability studies to: 1) assess the amounts of zinc-free and high-zinc LNS consumed by children during direct observation, 2) compare their mothers' sensory assessments of the respective products, and 3) review maternal reports of their child feeding experiences during more prolonged home feeding trials.

ELIGIBILITY:
Inclusion Criteria:

* Currently breast-feeding and consuming complementary foods for at least 30 d

Exclusion Criteria:

* Height-for-age and weight-for height Z-scores <-3 with respect to WHO growth standards
* Edema
* Diarrhea and other diseases that could interfere with food intake
* Severe systemic illness
* History of peanut allergy
* History of anaphylaxis/serious allergic reaction

Infants meeting these criteria and their mother's will be invited to participate

Ages: 9 Months to 15 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 36 (Actual)
Dates: Start 2009-07; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Amount of each type of LNS formulation consumed by young children | 3 days
Preference and detection of differences between LNS formulations among mothers | 3 days
Acceptability of feeding LNS to young children at home | 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth H. Brown, MD, Principal Investigator — University of California, Davis
Locations (1):
- Institut de Recherche en Sciences de la Santé, Bobo-Dioulasso, Burkina Faso

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Hess SY, Bado L, Aaron GJ, Ouedraogo JB, Zeilani M, Brown KH. Acceptability of zinc-fortified, lipid-based nutrient supplements (LNS) prepared for young children in Burkina Faso. Matern Child Nutr. 2011 Oct;7(4):357-67. doi: 10.1111/j.1740-8709.2010.00287.x. Epub 2010 Dec 15. PMID 21159124